CLINICAL TRIAL: NCT07260370
Title: The Difference of microRNA Signature(S) and Circulating Tumor Cells in Blood Among Cancer Patients Before and Afte Immunotherapy
Brief Title: The Difference of microRNA and Circulating Tumor Cells in Blood Among Cancer Patients With Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jason Chia-Hsun Hsieh, Professor Attending Physicians, Chang Gung Memorial Hospital
Other Study IDs: 201800596B0
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: microRNA; Circulating Tumor Cells; Immunotherapy
Keywords: Cancer; Plasma; Immunotherapy; microRNA; Circulating Tumor Cell
MeSH Terms: conditions — Neoplastic Cells, Circulating; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer for microRNA testing: The project will recruit 300 subjects who have been diagnosed with cancer by a physician and for whom the decision has been made to use immunotherapy. Blood samples will be collected before and after treatment (past pathological diagnostic tissues may also be reviewed as required for the study). The study will analyze the differences in the quantity of free microRNAs, the number of circulating tumor cells, and the differences in surface antigen expression in the subjects' blood, as well as the specific surface antigen expression status in the cancer tissues, and perform statistical analysis.

SUMMARY:
Among the currently important biomarkers, circulating tumor cells and microRNA (miRNA) have received significant attention. The latter, also translated as micro-ribonucleic acid, is a widely present ribonucleic acid (RNA) molecule in eukaryotes, approximately 21 to 23 nucleotides in length, which regulates the expression of other genes. miRNAs originate from RNAs that are transcribed from DNA but cannot be further translated into proteins (classified as non-coding RNA). miRNAs bind to target messenger RNA (mRNA), thereby inhibiting post-transcriptional gene expression, and play important roles in regulating gene expression, the cell cycle, and the timing of biological development.The project will recruit 300 subjects who have been diagnosed with cancer by a physician and for whom the decision has been made to use immunotherapy. Blood samples will be collected before and after treatment (past pathological diagnostic tissues may also be reviewed as required for the study). The study will analyze the differences in the quantity of free microRNAs, the number of circulating tumor cells, and the differences in surface antigen expression in the subjects' blood, as well as the specific surface antigen expression status in the cancer tissues, and perform statistical analysis.

DETAILED DESCRIPTION:
Among the currently important biomarkers, circulating tumor cells and microRNA (miRNA) have received significant attention. The latter, also translated as micro-ribonucleic acid, is a widely present ribonucleic acid (RNA) molecule in eukaryotes, approximately 21 to 23 nucleotides in length, which regulates the expression of other genes. miRNAs originate from RNAs that are transcribed from DNA but cannot be further translated into proteins (classified as non-coding RNA). miRNAs bind to target messenger RNA (mRNA), thereby inhibiting post-transcriptional gene expression, and play important roles in regulating gene expression, the cell cycle, and the timing of biological development.The project will recruit 300 subjects who have been diagnosed with cancer by a physician and for whom the decision has been made to use immunotherapy. Blood samples will be collected before and after treatment (past pathological diagnostic tissues may also be reviewed as required for the study). The study will analyze the differences in the quantity of free microRNAs, the number of circulating tumor cells, and the differences in surface antigen expression in the subjects' blood, as well as the specific surface antigen expression status in the cancer tissues, and perform statistical analysis.

For the trial, only two tubes of 10cc peripheral blood will be drawn (20cc total, using large purple-top collection tubes). Subjects will participate in a maximum of three blood draws for this trial (before immunotherapy, after immunotherapy, and during follow-up imaging).

Through drawing the patient's blood, extracting plasma, purifying microRNAs, and converting them into complementary deoxyribonucleic acid (cDNA)-in conjunction with cancer diagnostic materials (collected during past diagnoses, no new samples needed)-the miRSCanPanelChip™ platform will be utilized to screen and statistically analyze the quantity of free microRNAs in the plasma. Finally, the correlation between the RNA quantities, the number of circulating tumor cells, and the clinical treatment response will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged above 20 years.
2. A patient diagnosed with cancer with immunotherapy
3. Competent to give informed consent and agree to join the study.

Exclusion Criteria:

1. Aged < 20 years.
2. Refuse to join the study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The most crucial factor in preventing death for cancer patients is early diagnosis and the detection of recurrence.The project will recruit 300 subjects who have been diagnosed with cancer by a physician and for whom the decision has been made to use immunotherapy. Blood samples will be collected before and after treatment. The study will analyze the differences in the quantity of free microRNAs, the number of circulating tumor cells, and the differences in surface antigen expression in the subjects' blood, as well as the specific surface antigen expression status in the cancer tissues, and perform statistical analysis
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
counting of Circulating Tumor Cells | baseline,pre-iprocedure
  The study will do the counting of circulating tumor cells in the participants with immunotherapy.
counting of Circulating Tumor Cells | 3 month, during procedure
  The study will do the counting of circulating tumor cells in the participants with immunotherapy.
counting of Circulating Tumor Cells | 6 month
  The study will do the counting of circulating tumor cells in the participants with immunotherapy.

SECONDARY OUTCOMES:
microRNAs sequence | baseline,pre-iprocedure
  The study will analyze the differences in the quantity of free microRNAs
microRNAs sequence | 3 month, during procedure
  The study will analyze the differences in the quantity of free microRNAs
microRNAs sequence | 6 month
  The study will analyze the differences in the quantity of free microRNAs

OTHER OUTCOMES:
Treatment response | 3 month, during procedure
  Record the response after immuntherapy
Treatment response | 6 month
  Record the response after immuntherapy

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, PhD, Principal Investigator — Division of Oncology, Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan